CLINICAL TRIAL: NCT05247671
Title: Evaluation of the Effect of Genetic Polymorphisms in ERCC1 and OCT2 on the Occurrence and Severity of Cisplatin-induced Nephrotoxicity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: PG study on cisplatin
Record Dates: First submitted 2021-12-10; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-11

CONDITIONS: Cisplatin Adverse Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Case: All eligible patients will be recruited to the study and will be assessed for SNPs in both ERCC1 and OCT2 and their association with cisplatin-induced nephrotoxicity through the measurement of cystatin C before taking cisplatin and after receiving the second cycle of cisplatin.
  Interventions: Genetic: ERCC1; Genetic: OCT2

INTERVENTIONS:
Genetic: ERCC1 — ERCC1 is a rate-limiting enzyme in the nucleotide excision repair pathway that is known to repair cisplatin-induced DNA damage. Polymorphisms in ERCC1 are known to affect response to cisplatin treatment. A mechanism explaining the effect of the ERCC1 polymorphism on the kidney may be that the homozygous carriers of this rs3212986 allele might have a greater capacity to repair cisplatin-induced DNA damage in their kidney epithelia, and thus would be more resistant to cisplatin-induced nephrotoxicity
Genetic: OCT2 — OCT2 is expressed on the basolateral membrane of Proximal Tubular Epithelial Cell (PTEC) and plays a central role in cisplatin uptake into tubular cells. Genetic variants in the cisplatin uptake transporter OCT2 showed association with the preservation of kidney function. Patients with the CT genotype in OCT2 polymorphism rs596881 exhibited positive changes in eGFR compared to individuals with the wild type CC genotype

SUMMARY:
Approximately one-third of all patients treated with cisplatin develop renal dysfunction after a single dosage of cisplatin. Germline genetic polymorphisms may cause variations in cisplatin pharmacokinetics and in the ability of epithelial kidney cells to take up cisplatin and repair cisplatin-induced Deoxyribonucleic Acid (DNA) damage. Knowledge concerning which genotypes are associated with cisplatin-induced nephrotoxicity may help to identify at-risk patients and initiate strategies, such as using lower or fractionated cisplatin doses or avoiding cisplatin altogether, to prevent Acute Kidney Injury (AKI).

DETAILED DESCRIPTION:
Approximately one-third of all patients treated with cisplatin develop renal dysfunction after a single dosage of cisplatin. Germline genetic polymorphisms may cause variations in cisplatin pharmacokinetics and in the ability of epithelial kidney cells to take up cisplatin and repair cisplatin-induced DNA damage. Knowledge concerning which genotypes are associated with cisplatin-induced nephrotoxicity may help to identify at-risk patients and initiate strategies, such as using lower or fractionated cisplatin doses or avoiding cisplatin altogether, to prevent AKI.

Patient written informed consent will be taken prior to study conductance

1. Full laboratory evaluation before and after cisplatin administration including:

   (Complete Blood Count) CBC, liver and renal functions. glomerular filtration rate (GFR), and estimated glomerular filtration rate (eGFR) Serum electrolytes. Marker of nephrotoxicity: Cystatin C.
2. Sample Collection and single nucleotide polymorphism (SNP) Genotyping:

Venous blood (2 mL) will be collected from each subject into tubes containing 50 mmol of Ethylenediamine tetraacetic acid (EDTA) per liter and genomic DNA will be isolated with the GeneJET Whole Blood Genomic DNA purification Mini kit, according to manufacturer's instructions. Polymorphisms will be assessed using the TaqMan based real-time polymerase chain reaction (PCR) assay.

This study aims to assess the influence of single nucleotide polymorphisms in the DNA repair gene Excision Repair Cross Complementation group 1 (ERCC1) and Cisplatin uptake transporter gene Organic Cation Transporter 2 (OCT2) on cisplatin-induced nephrotoxicity by assessment of the following:

1. Occurrence of nephrotoxicity.
2. Degree of renal impairment.
3. Changes in traditional and novel protein biomarkers for AKI.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged >18 years receiving cisplatin-containing chemotherapy.
* A Cisplatin dose starting from 75 mg/m2
* Various cancer types
* No history of organ transplantation or kidney dialysis.
* Patients with normal renal function

Exclusion Criteria:

* Co-administration of ifosfamide with cisplatin, because of the known risk of nephrotoxicity.
* Pregnant or lactation.
* Infection with the human immunodeficiency virus (HIV).
* Prior administration of cisplatin.
* Intraperitoneal chemotherapy.
* Inadequate liver function (bilirubin > 1.5 times upper normal limit (UNL) and alanine transaminase (ALT) or aspartate transaminase (AST) > 3.0 UNL or up to 5.0 UNL in the presence of hepatic metastases).
* Inadequate renal function (creatinine > 1.25 times UNL, creatinine clearance < 50 mL/min).
* Serious comorbid systemic disorder incompatible with the study (uncontrolled diabetes mellitus (DM) or hypertension (HTN), myocardial infarction within the last 6 months).
* Patients diagnosed with kidney cancer.
* Exposure to any nephrotoxic drugs or agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males or females aged >18 years receiving cisplatin-containing chemotherapy presenting to the Department of Oncology, faculty of medicine, Ain Shams University will be assessed for eligibility according to the inclusion & exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2022-08-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Serum Creatinine | Change from baseline at the end of cycle 1 (each cycle is 28 days)
  available in patient profile
Serum Creatinine | Change from baseline at the end of cycle 2 (each cycle is 28 days)
  available in patient profile

SECONDARY OUTCOMES:
cystatin c | Change from baseline at the end of cycle 2 (each cycle is 28 days)
  measured by Human cystatin C ELISA kit

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Elwakeel, Study Director — Head of Clinical Department, Faculty of Pharmacy, Ain Shams University
Locations (1):
- Faculty of medicine, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided